CLINICAL TRIAL: NCT05863780
Title: Comparison of Flexor Retinaculum Stretch and Carpal Mobilizations in Patients With Carpal Tunnel Syndrome on Pain, ROM and Functional Status
Brief Title: Comparison of Flexor Retinaculum Stretch and Carpal Mobilizations in Patients With Carpal Tunnel Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/RCRS/REC/01317
Record Dates: First submitted 2023-02-20; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: median neuropathy; thenar muscle atrophy; compression neuropathy; flexor retinaculum
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy; Tomaculous neuropathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carpal bone mobilization (Experimental): Carpal bone mobilization will be done
  Interventions: Other: Carpal bone mobilization
- Flexor retinaculum stretch (Experimental): Flexor retinaculum stretch will be given.
  Interventions: Other: Flexor retinaculum stretch
- Carpal bone mobilization and flexor retinaculum stretch (Experimental): Carpal bone mobilization and flexor retinaculum stretch will be given together
  Interventions: Other: Carpal bone mobilization and flexor retinaculum stretch

INTERVENTIONS:
Other: Carpal bone mobilization — Carpal bone mobilization 5 repetition/1 set lasted for 15 secs followed by 10 secs of rest- 3 sessions on alternate days per week for 04 weeks.
  Total of 12 sessions will be given, each consisting of 45 mins.
  Arms: Carpal bone mobilization
Other: Flexor retinaculum stretch — Flexor retinaculum stretch 5 repetitions/ 1 set held for 60 secs at a time,-3 sessions on alternate days per week for 04 weeks.
  Total of 12 sessions will be given, each consisting of 45 mins.
  Arms: Flexor retinaculum stretch
Other: Carpal bone mobilization and flexor retinaculum stretch — 1. Carpal bone mobilization 5 repetition/1 set lasted for 15 secs followed by 10 secs of rest.3 sessions on alternate days per week for 04 weeks.
  2. Flexor retinaculum stretch 5 repetitions/ 1 set held for 60 secs at a time-3 sessions on alternate days per week for 04 weeks.
  Total of 12 sessions will be given, each consisting of 45 mins.
  Arms: Carpal bone mobilization and flexor retinaculum stretch

SUMMARY:
Comparison of flexor retinaculum stretch and carpal mobilizations in carpal tunnel syndrome patients.

DETAILED DESCRIPTION:
* Carpal Bones Mobilization tends to improve the symptoms of carpal tunnel syndrome.
* Manual stretching of the flexor retinaculum effective in CTS patients.
* As there are no studies available to compare the effectiveness of flexor retinaculum stretch and carpal bone mobilization for the treatment of CTS, hence the purpose of this study is to find the effectiveness of carpal bone mobilization and flexor retinaculum stretch in improving Pain, ROM and Functional Status in patient with CTS.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age between 18-40 years
* Unilateral CTS
* Already diagnosed patients of CTS.

Exclusion Criteria:

* Fracture of wrist
* Dislocation
* Congenital abnormalities
* Rheumatoid arthritis
* Osteoarthritis
* Liver failure
* Pregnancy
* Bilateral CTS
* Systemic neurological condition e.g.: GB syndrome, multiple sclerosis.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4th week
  Changes from baseline. NPRS is an 11 point numeric scale scored from 0-10. The maximum pain value is 10. 0 means no pain whereas 10 means most intense pain imaginable
Boston Carpal Tunnel Questionnaire (BCTQ) scale (SSS, FSS) | 4th week
  Changes from baseline. The Boston Carpal Tunnel Score is a patient-reported questionnaire that examines symptom severity and overall functional status. It has two subscales.
  1. The Symptom Severity Scale (SSS) with 11 questions is scored on a Likert scale from 1-5 where 1 means no symptom and 5 means most severe symptom. The maximum score is 55.
  2. The Functional Status Scale (FSS) with 8 questions is scored from 1-5 with 1 as no difficulty and 5 as "cannot do at all due to hand or wrist symptoms". The maximum score is 40.
6-item CTS symptoms scale (CTS-6) | 4th week
  Changes from baseline.The CTS-6 was scored with conventional scoring (similar to that used for the 11-item symptom severity scale) each item was scored on a scale of 1 (no symptom) to 5 (most severe symptom).
ROM wrist flexion | 4th week
  Changes from baseline ROM range of motion of wrist flexion was taken by using Goniometer
ROM wrist extenion | 4th week
  Changes from baseline ROM range of motion of wrist extension was taken by using Goniometer
ROM radial deviation | 4th week
  Changes from baseline ROM range of motion of radial deviation was taken by using Goniometer
ROM ulnar deviation | 4th week
  Changes from baseline ROM range of motion of ulnar deviation was taken by using Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Rawal Institute of Health Sciences, Rawalpindi, Punjab Province
  - Islamabad physiotherapy rehabilitation centre, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No